CLINICAL TRIAL: NCT06710730
Title: Joy in Work, Resilience Capacity, and Patient Safety Culture Among Healthcare Professionals In-hospital
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Irene Lie, Professor. Senior researcher, Oslo University Hospital
Other Study IDs: 2024/22563
Record Dates: First submitted 2024-11-22; First posted 2024-11-29 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-11

CONDITIONS: No Condition is the Focus of the Study
Keywords: Joy in Work. Resilience Capacity. Patient Safety Culture. Health care professionals. Inhospital.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Health care professionals working at Department of Cardiothoracic surgery: Longitudinal 3-year study. Data collection 2024 - 2026

SUMMARY:
In this project, the investigators will investigate three important factors to optimize working conditions and patient safety: Joy in Work, Resilience Capacity, and Patient safety culture using both questionnaires and focus group interviews.

DETAILED DESCRIPTION:
Already in 2021, the Norwegian Patient Safety Conference 'In Safe Hands 24-7' focused on adaptability: "How can health care professionals learn from what goes well?" Working to be excellent, identifying areas for improvement, and succeeding in a continuous improvement process. A solid patient safety culture requires competent and adaptable health care professionals, leaders, and health care systems. Joy in work is the experiential factor that revolves around opportunities for personal development, influencing one's own work, having individual contributions valued, and feeling like a meaningful part of the community.

This project spans three years-before (2024), during (2025), and after (2026) the physical co-location of Department of Cardiothoracic Surgery at Oslo university hospital. Four-hundred (n=400) health care professionals are working at Department of Cardiothoracic surgery, Oslo University Hospital, Norway and are eligible to be included in the study.

Health care professionals view of Joy in Work, Resilience Capacity, and Patient safety culture will be described using three international questionnaires. It is within the scope of the study to perform sub-analysis due to sub-categories of the questionnaires. Analysis across the questionnaires will be performed.

Furthermore, the three terms Joy in Work, Resilience Capacity, and Patient safety culture will be explored by approximately 10 % of the four-hundred (n=40) health care professionals in 5-6 focus group interviews, in 2024, 2025 and 2026..

ELIGIBILITY:
Inclusion Criteria:

* Health care professionals working at Department of Cardiothoracic Surgery

Exclusion Criteria:

* Not able to understand the Norwegian questionnaires

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — All kind of gender-
Study Population: All health care professionals working at Department of Cardiothoracic Surgery November/December 2024, 2025 and 2026. 400 employees x 3 years, a total of 1200 possible respondents.
  This is a descriptive and exploratory study (i.e., no priority given to a specific hypothesis). No relevant studies available to estimate the number of participants needed in this study. To detect medium effect sizes (Cohen's d=0.5) between groups, need to include a total of 172 participants, considering a type I error rate of 5% and a power of 90%. Two-sided t-test were used as the basis for this calculation. In addition, we aim to investigate factors associated with job satisfaction, resilience capacity, or patient safety culture. A sample of 147 participants would be sufficient to detect a small to medium effect size (f2=0.08) with 90 % power and a type I error of 5% in a multiple linear regression model with ten predictor variables. Sufficient power for analyzing subscales/subgroups, aim include 400.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2027-03-25 (Estimated); Study Completion 2027-03-25 (Estimated)

PRIMARY OUTCOMES:
Describe Joy in Work among health care professionals at Department of Cardiothoracic surgery | December 2024, 2025 and 2026
  Health care professionals working at Department of Cardiothoracic surgery in November/December 2024-2026 will be invited to participate in the longitudinal 3-year study.
  Sub analysis will be performed for sub scales/sub-themes of the questionnaires: Joy of Work (39 questions)
  This descriptive study is categorized as anonymous by the hospitals Data Protection Officer. Electronic web based questionnaire will be forwarded to all health care professionals at Department of Cardiothoracic surgery

SECONDARY OUTCOMES:
Describe Resilience Capacity among health care professionals at Department of Cardiothoracic surgery | November/December 2024-2026
  Health care professionals working at Department of Cardiothoracic surgery in November/December 2024-2026 will be invited to participate in the longitudinal 3-year study.
  Sub analysis will be performed for sub scales/sub-themes of the questionnaire Resilience Capacity (33 questions)
Describe Patient Safety Culture among health care professionals at Department of Cardiothoracic surgery | November/December 2024-2026
  Health care professionals working at Department of Cardiothoracic surgery in November/December 2024-2026 will be invited to participate in the longitudinal 3-year study. Sub analysis will be performed for sub scales/sub-themes of the questionnaire Patients safety culture (HSOPS 2.0) (36 questions)

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Oslo University Hospital, Oslo, Oslo County
  - Department of Cardiothoracic surgery, Division on Cardiovascular and Pulmonary Diseases, Oslo University hospital, Oslo

IPD SHARING:
Plan to Share IPD: No
Not included in the informed consent to the respondents